CLINICAL TRIAL: NCT04601675
Title: Randomized Study on Diabetic Macular Edema Patients Receiving Ranibizumab and Dexamethasone or Ranibizumab Only.
Brief Title: Diabetic Macular Edema (DME) Treatment With Ranibizumab and Dexamethasone or Ranibizumab Only.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: He Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ME-230620
Record Dates: First submitted 2020-10-20; First posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-06

CONDITIONS: Macular Edema
MeSH Terms: conditions — Macular Edema | interventions — Ranibizumab; Calcium Dobesilate

STUDY DESIGN:
Intervention Model Description: Drug: Ozurdex intravitreal steroid Other Name: Dexamethasone Intravitreal Implant Drug: Bevacizumab antiVEGF Other Name: Avastin
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetic ME: Ranibizumab and intravitreal Dexamethasone (Experimental): Participants with diabetic macular edema will receive a combination of Ranibizumab and intravitreal Dexamethasone
  Interventions: Drug: Ranibizumab Ophthalmic and Intravitreal Dexamethasone
- Diabetic ME: Ranibizumab (Active Comparator): Participants with diabetic macular edema (ME) will receive Ranibizumab only.
  Interventions: Drug: Ranibizumab Ophthalmic only

INTERVENTIONS:
Drug: Ranibizumab Ophthalmic and Intravitreal Dexamethasone — Pro re nata patients with macula edema due to diabetes will receive Ranibizumab. Group A will continue to receive Ranibizumab depending on their clinical status of macular edema
  Other Names: Lucentis®; Ozurdex®
  Arms: Diabetic ME: Ranibizumab and intravitreal Dexamethasone
Drug: Ranibizumab Ophthalmic only — Group B will initially receive intravitreal Dexamethasone and Ranibizumab and then depending on their clinical status of macular edema, Ranibizumab will be injected.
  Other Names: Lucentis®
  Arms: Diabetic ME: Ranibizumab

SUMMARY:
The aim of this study is to evaluate the visual outcome and prognostic factors after intraocular injections of Ranibizumab or combination of Ranibizumab And Dexamethasone under pro re nata treatment regimen for Diabetic Macular Edema patients.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the clinical outcome after intraocular injections of Ranibizumab or combination of Ranibizumab and Dexamethasone under pro re nata treatment regimen for the patients with Diabetic Macular Edema patients. Mean change of logarithm of the minimal angle of resolution (logMAR) visual acuity (VA), central foveal thickness (CFT), contrast sensitivity (CS) as well as predictive factors including best-corrected visual acuity (BCVA), vision related questionnaires and various other ocular parameters will be assessed.

ELIGIBILITY:
Inclusion Criteria:

Patients with diabetic retinopathy and centre involving DMO, as determined by using spectral domain optical coherence tomography (SD-OCT), in one or both eyes with:

1. Central retinal subfield thickness of > 300 but < 400 microns as determined by SD-OCT due to diabetic macular oedema OR
2. Central retinal subfield thickness of < 300 microns provided that intraretinal and/or subretinal fluid is present in the central subfield (central 1 mm) related to diabetic macular oedema AND
3. Visual acuity of > 24 Early Treatment Diabetic Retinopathy Study (ETDRS) letters (Snellen equivalent > 20/320)
4. Amenable to laser treatment, as judged by the treating ophthalmologist
5. Over 18 years of age

Exclusion Criteria:

Eyes of patients will not be included in the study if:

1. The macular oedema is due to causes other than diabetic macular oedema such as epiretinal membrane, vitreomacular traction, vein occlusion, or others
2. The eye is ineligible for macular laser treatment, as judged by the treating ophthalmologist
3. The eye has DMO and central subfield retinal thickness (CST) of > 400 microns.
4. The eye has activeA proliferative diabetic retinopathy (PDR) requiring treatment.
5. The eye has received intravitreal Anti- Vascular Endothelical Growth Factor (Anti-VEGF) therapy within the previous two months.
6. The eye has received macular laser treatment within the previous 12 months.
7. The eye has received intravitreal injection of steroids.
8. The eye has received cataract surgery within the previous six weeks
9. The eye has received panretinal photocoagulation within the previous 3 months
10. Patients on pioglitazone and the drug cannot be stopped 3 months prior to entering into the trial and for the duration of the study
11. The patient has chronic renal failure requiring dialysis or kidney transplant
12. The patient has any other condition that in the opinion of the investigator would preclude participation in the study (such as unstable medical status or severe disease that would make it difficult for the patient to be able to complete the study)
13. The patient has very poor glycemic control and started intensive therapy within the previous 3 months
14. The patient will use an investigational drug during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-10-31 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-09-17 (Estimated)

PRIMARY OUTCOMES:
Mean change in monocular BCVA in the treatment eye | Baseline, 1 week, 1month, 2 months, 3 months, and 6 months.
  Monocular BCVA in the treatment eye is assessed by using ETDRS visual acuity charts at 4 meters at baseline (pre-treatment) and 1 week, 1month, 2 months, 3 months, and 6 months after treatment.
Mean change in binocular BCVA | Baseline, 1 week, 1month, 2 months, 3 months, and 6 months.
  Binocular BCVA is assessed by using ETDRS visual acuity charts at 4 meters at baseline (pre-treatment) and 1 week, 1month, 2 months, 3 months, and 6 months after treatment.

SECONDARY OUTCOMES:
Mean change in central subfield retinal thickness | Baseline, 1 week, 1month, 2 months, 3 months, and 6 months.
  Mean change in central subfield retinal thickness in the study eye, as determined by spectral domain optical coherence tomography (OCT), from baseline to 6 months.
Change in Humphrey 10-2 visual field in the treatment eye | Baseline, 1 week, 1 month, 2 months, 3 months, and 6 months.
  Mean deviation (MD) of the Humphrey 10-2 visual field is assessed by a Humphrey 10-2 visual field test at baseline, 1 week, 1month, 2 months, 3 months, and 6 months.
People meeting driving standards | Baseline, 1 week, 1 month, 2 months, 3 months, and 6 months.
  Percentage (%) of people meeting driving standards is assessed by an Esterman binocular visual field test at baseline and and 6 months.
Mean change in NEI VFQ25 | Baseline, 1 week, 1 month, 2 months, 3 months, and 6 months.
  Scores from NEI VFQ25 questionnaire will be assessed and compared at baseline, 1 week, 1 month, 2 months, 3 months, and 6 months.
Mean change in EQ-5D 5L | Baseline, 1 week, 1 month, 2 months, 3 months, and 6 months.
  Scores from EQ-5D 5L questionnaire will be assessed and compared at baseline, 1 week, 1 month, 2 months, 3 months, and 6 months.
Mean change in VisQoL scores | Baseline, 1 week, 1 month, 2 months, 3 months, and 6 months.
  Scores from VisQoL questionnaire will be assessed and compared at baseline, 1 week, 1 month, 2 months, 3 months, and 6 months.
Mean change in wavefront aberrations | Baseline, 1 week, 1 month, 2 months, 3 months, and 6 months.
  Mean deviation (MD) of wavefront aberrations is assessed by Nidek OPD Scan III test at baseline, 1 week, 1month, 2 months, 3 months, and 6 months.
Mean change in ocular surface and tear-film | Baseline, 1 week, 1 month, 2 months, 3 months, and 6 months.
  Mean deviation (MD) of ocular surface and tear-film parameters is assessed by Oculus Keratographer test at baseline, 1 week, 1month, 2 months, 3 months, and 6 months.
Mean change in vessel density | Baseline, 1 week, 1 month, 2 months, 3 months, and 6 months.
  Mean deviation (MD) of vessel density is assessed by Spectralis OCT2, Heidelberg-Engineering test at baseline, 1 week, 1month, 2 months, 3 months, and 6 months.
Side effects | 1 week, 1 month, 2 months, 3 months, and 6 months.
  Side effects are measured by a review of the participant's medical and ophthalmic history.
Use of additional treatments (including laser) | 1 week, 1 month, 2 months, 3 months, and 6 months.
  Use of additional treatments (including laser) is assessed by the treating ophthalmologist

CONTACTS AND LOCATIONS:
Overall Officials: Wei He, M.D., Ph.D., Study Chair — He Eye Specialist Hospital, Shenyang.; Jun Li, M.D., Ph.D., Principal Investigator — He Eye Specialist Hospital, Shenyang.; Emmanuel E Pazo, M.D., Ph.D., Study Director — He Eye Specialist Hospital, Shenyang.
Locations (1):
- He Eye Specialist Hospital, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No